CLINICAL TRIAL: NCT04414774
Title: Assessing the Effectiveness of a CBT-based App in Reducing Suicidal Ideation: An Open Randomized Study
Brief Title: Assessing the Effectiveness of a CBT-based App in Reducing Suicidal Ideation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahak Yariv (Other)
Collaborators: Interdisciplinary Center Herzliya (Other)
Responsible Party: Sponsor-Investigator, Shahak Yariv, Senior physician in mental health care and neuromodulation service manager, HaEmek Medical Center, Israel
Organization: HaEmek Medical Center, Israel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMC-0108-19; 201912001 (Other: Ministry of Health Israel)
Record Dates: First submitted 2020-05-20; First posted 2020-06-04 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Suicide Ideation
Keywords: Suicide ideation; Mental pain; Mobile app; Application

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the control or experimental group. The experimental group will immediately start using the GGSI app, for a period of 15 days (T1), while the control group waits. After 15 days (T2) the experimental group ceases its use of the app. At the same time, the control group will start its 15-days usage of the app. The end of these 15 days is marked T3.
Masking Description: There is no masking in this research, since the research team needs to know what stage the subjects are in in order to conduct the study. Due to ethical considerations, the subjects are aware that the purpose of the app is to reduce mental distress and suicidal ideation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- using app first (Experimental): The experimental group will immediately start using the GGSI app, for a period of 15 days (T1). After 15 days (T2) the experimental group ceases its use of the app. The end of this period is marked T3. The research team will contact the experimental group on T1, T2 and T3 in order to fill out questionnaires regarding suicide ideation and related risk factors.
  Interventions: Device: GG-Suicide-Ideation
- waiting list (Active Comparator): During the first 15 days, the control group is inactive (T1). After 15 days (T2) the control group will start using GGSI app for additional 15 days (T3). Participants will fill questionnaires about suicide ideation and related risk factors three time during the study on: T1, T2 and T3.
  Interventions: Device: GG-Suicide-Ideation

INTERVENTIONS:
Device: GG-Suicide-Ideation — GG-Suicide-Ideation (GGSI) is a mobile application, consisting of 55 stages. The content of each stage is a list of statements representing core themes, that were found in research and clinical practice to be related to suicide ideation. These are, for example, hopelessness, helplessness, thwarted belongingness, perceived burdensomeness, low self-esteem, tolerance of mental pain, and more. On each stage, several statements are presented on screen, one at a time. The statements express adaptive or maladaptive thinking in the specific core theme of that stage. In case the statement is positive and adaptive, the user needs to drag the statement downwards, towards him. In case the statement is negative and maladaptive, the user needs to drag the statement upwards, away from him. The user advances in stages - three stages per day.

SUMMARY:
The aim of this study is to empirically assess the utility of GG-Suicide-Ideation (GGSI), a theory-based mobile application for the prevention of suicide ideation. GGSI is based on principles of Cognitive Behavioral Therapy (CBT), which have been found to be an effective treatment for decreasing suicide risk.

In this study half of the participants (i.e. the experiment group) will start an immediate use of GGSI for a period of 15 days. The other half of the participants (i.e. the control group) will be 'on hold' during the first 15 days, after which they will commence use of GGSI for an additional 15 days.

All participants will complete questionnaires regarding suicide ideation and related risk factors three times during the study: at the beginning of the study (baseline), after 15 days from the beginning of study and after 30 days from the beginning of study.

The investigators hypothesized that in the experimental group, after 15 days of using GGSI app there will be a substantial decrease in the level of suicide ideation and associate risk factors, compared to the control group. If this hypothesis is met, the investigators will examine if the decrease in said measures in the experimental group will maintain after 15 days of follow up. In addition, the investigators hypothesized that in the control group there will be a significant decrease in suicide ideation and related risk factors after 15 days of using GGSI.

DETAILED DESCRIPTION:
Introduction:

Suicide is a leading cause of death in many countries. One of the major risk factors of suicide is suicide ideation. Different theories describe the developing path and the association between suicide ideation, suicide attempts, and, eventually, suicide. Given the existing continuum between suicide ideation, suicidal behavior, and suicide, an effective suicide prevention strategy may focus on reducing suicide ideation.

Suicide ideation is an expression of distress and is associated with various risk factors. Among risk factors are depression, mental pain, tolerance of mental pain, hopelessness and helplessness, low self-esteem, thwarted belongingness and perceived burdensomeness.

Suicide ideation and cognition: Historical review on the association between cognition and suicide ideation indicates that there are maladaptive thinking patterns ("cognitive distortions") that exist substantially among suicidal individuals, compared to non-suicidal subjects. Furthermore, David Lester, a well-known researcher in the field of suicidality, examined seven theory-based risk factors for suicide behavior and suggested that they may be considered as the maladaptive cognitive distortions which stand in the core of suicide behavior. The risk factors for suicide ideation, which are mentioned in the head of this paper, are very much congruent to those suggested by Lester, and may be considered as part of the maladaptive thinking patterns that form the basis of suicide ideation and behavior.

Cognitive change as an effective intervention for decreasing suicide ideation: One of the renowned treatments which put a great emphasis on changing maladaptive thinking patterns in order to alleviate the psychological pain of the patient is Cognitive Behavioral Therapy (CBT). CBT is an effective treatment for decreasing suicide risk. CBT is based on the theoretical assumption that the way people think about and interpret life events determines their emotional and behavioral responses to those events. This model suggests that cognitive distortions (repeated distortions in thinking and interpreting reality) are imperative to the formation of suicide thoughts and behavior.

Cognitive-behavioral therapies have been found effective for preventing suicide. After coping with the acute suicide crisis, the treatment emphasizes changing maladaptive schemes and thoughts. According to this and to other findings, it can be assumed that cognitive adaptation is a significant change agent in the reduction of suicide ideation and behavior. Furthermore, it can be said that an intervention designed to challenge dysfunctional thoughts and create accessible adaptive thoughts, in areas previously found to predispose suicidal thoughts, can promote the reduction of suicide ideation.

One way to make this kind of intervention accessible to the general public is through an application. Today there is more awareness to the fact that many individuals who require care do not receive treatment. An application may be a possible solution to overcome this clinical gap and alleviate the suffering of individuals with suicide ideation in the general public. Moreover, an application delivered by smartphones has excellent potential to be acceptable by the user due to its availability, low effort expectancy, and high hedonic motivation.

Suicide prevention and mobile applications: The empirical literature shows an increasing number of mobile applications focusing on preventing suicide. Some of the existing apps contain elements that have been found to be effective for suicide prevention. Most of the apps designated for suicidal crisis and contain multiple interventions. Two applications that were empirically assessed failed to show a substantial decrease in suicide ideation following usage. However, it should be noted that these studies employed a small sample size, and therefore lack statistical power.

The current study: The aim of this study is to empirically assess the utility of GG-Suicide-Ideation (GGSI), a theory-based mobile application for the prevention of suicide ideation. GGSI is based on principles of CBT, which have been found to be an effective treatment for suicidality. Particularly GGSI aims to challenge suicidal maladaptive thoughts and to increase accessibility of adaptive thinking patterns in relevant domains. All of this being done by a daily practice which is delivered in a game-like manner. Moreover, GGSI provides a missing element in the domain of suicide prevention apps: as far as the investigators know, there is no app or internet program for suicide prevention, which is delivered in a game-like manner. In addition, GGSI is designated for daily use, as opposed to most apps, which target suicidal crisis periods specifically. Moreover, the format which GGSI is based on was tested on OCD (Obsessive-Compulsive Disorder) symptoms and found effective.

Considering all of the above, the investigators hypothesize that in the experimental group after 15 days of using GGSI app, there will be a substantial decrease in the level of suicide ideation, mental pain, depression and in measures related to suicidal maladaptive thinking patterns (i.e. tolerance of mental pain, hopelessness, helplessness, low self-esteem, thwarted belongingness and perceived burdensomeness) versus the control group which are on hold for GGSI usage. If this hypothesis will be met, the investigators will examine if the decrease in these measures in the experimental group sustain after 15 days of follow up. In addition, the investigators hypothesize that in the control group there will be a significant decrease in the mentioned measures after 15 days of using GGSI.

Methods

Participant: Participation in the study will be offered to all patients present in the adult-depression unit of the outpatient clinic of Medical Center Ha'emek. Participant recruitment will be done by the treating psychiatrist, who will examine the participants suitability for the study by inclusion and exclusion criteria. Participation in the study will be offered to patients as an adjunct to their proposed psychiatric and psychotherapeutic treatment. The study was approved by the IRB committee.

Sample and power analysis: Power analysis was conducted using G*Power. For α = 0.05, the statistical power is 0.80 and the effect size is medium (f=0.25). Hence, 128 subjects are required for the requested analysis, and this number of participants will be recruited.

Study design: Participants will sign a consent form. The course of the study will be explained to all participant. In the experimental group, after filling out the relevant questionnaires, participants will be explained how to download the GGSI app to their mobile phone, and that they will need to use the app once a day for 15 days. In the control group, participants will be explained that they are now filling out questionnaires and in 15 days they will be invited to another meeting to fill out additional questionnaires and receive the app. The research team will contact participants via a phone call at the following time points: first, seven days after they received the app, the research team will remind and encourage the participants to continue using the GGSI app every day. Second, each time filling out questionnaires is needed (except from when participants fill out questionnaires in the outpatient clinic, see above) the research team will call the subjects, conduct a suicide risk assessment according to the Colombia suicide severity rating scale (C-SSRS). They will also ask participants to fill out questionnaires via the app or a link sent to their phone. Third, after the 15 days app usage period, the participants will be asked to remove the GGSI app from their phone.

Suggested Statistical analysis: As been done before in research on an application with similar interface and with similar study design (waiting list control add on), a series of repeated Measure ANOVA with Bonferroni adjustments, will be calculated in order to asses pre-post scores in both study groups.

Ethical considerations:

The aim of GGSI app is to reduce emotional stress. In any case where participants feel that using the app cause them distress, they can stop the usage in any given time. If the participant requires additional assistance or support, that will be provided to them by the research team. Along the study period, in any case where suicide risk immerges from the questionnaire scores or from subject suicide risk assessment or from any complaint done by a participant, an initial assessment will be made. In case of actual suicide risk, the relevant participant will be referred to suicide risk assessment by the clinic staff or to the emergency room, and their treatment will be transferred to Dr. Yariv Shahak, manager of the depression clinic.

Privacy and information security:

When downloading the app, the information needed for registration is the participant's gender and age. The app does not receive accurate information about the location of the mobile device. While subjects use the app, its output is transmitted to a secure server. The information on the server is stored anonymously, and with no identifying details. The app output will be deleted at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speakers
* Subjects at a low suicide risk only (see note below).
* Patients who suffered from passive suicide ideation in the past two weeks.
* Participants must have a mobile phone capable of supporting the GGSI app.

Exclusion Criteria:

* Patients at moderate to high suicide risk, as determined by The Columbia- Suicide Severity Rating Scale (C-SSRC; Posner et al., 2011)
* Patients diagnosed with psychosis or autism, and drug users.
* Patients who are admitted to the ER, or are hospitalized in the psychiatric wards.

  * Suicide risk will be determined by The Columbia- Suicide Severity Rating Scale (C-SSRC; Posner et al., 2011). In accordance with this scale, we defined at a low suicide risk patients who have suicide ideation but without a method of execution, suicide intention, or suicide plan. At moderate to high suicide risk we defined patients who indorse suicide ideation with a method of execution and\or suicide intention and\or suicide plan.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Adult Suicide Ideation Questionnaire (ASIQ) at Day 15. | Baseline and Day 15.
  Frequency of suicide ideation in the past two weeks will be assessed using a self-report questionnaire (Adult Suicide Ideation Questionnaire (ASIQ) ; Reynolds, 1991). The questionnaire contains 25 items. Each item is scored on a scale of 0-6, yielding a total score of between 0-150. Higher score indicates a greater frequency and severity of suicide ideation. Change= (Day 15 score - baseline score).
Change from Day 15 in Adult Suicide Ideation Questionnaire (ASIQ) at Day 30. | Day 15 and Day 30.
  Frequency of suicide ideation in the past two weeks will be assessed using a self-report questionnaire (Adult Suicide Ideation Questionnaire (ASIQ) ; Reynolds, 1991). The questionnaire contains 25 items. Each item is scored on a scale of 0-6, yielding a total score of between 0-150. Higher score indicates a greater frequency and severity of suicide ideation. Change= (Day 30 score - Day 15 score).
Change from Baseline in Quick Inventory of Depressive Symptomatology Questionnaire (QIDS) at Day 15. | Baseline and Day 15.
  Severity of depressive symptoms in the past week will be assessed using a self-report questionnaire (Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR16); Rush et al., 2003). The questionnaire contains 16 items. Each item is scored on a scale of 0-3. Higher score indicates a greater number and severity of depressive symptoms. Change= (Day 15 score - baseline score).
Change from Day 15 in Quick Inventory of Depressive Symptomatology Questionnaire (QIDS) at Day 30. | Day 15 and Day 30.
  Severity of depressive symptoms in the past week will be assessed using a self-report questionnaire (Quick Inventory of Depressive Symptomatology Self-Report (QIDS-SR16); Rush et al., 2003). The questionnaire contains 16 items. Each item is scored on a scale of 0-3. Higher score indicates a greater number and severity of depressive symptoms. Change= (Day 30 score - Day 15 score).
Change from Baseline in Orbach and Mikulincer Mental Pain scale (OMMPI) at Day 15. | Baseline and Day 15.
  The experience of mental pain will be assessed using a self-report questionnaire (OMMPI; Orbach, Mikulincer, Sirota & Gilboa-Schechtman, 2003). The questionnaire contains 44 items. Each item is scored on a scale of 1-5, yielding a total score of between 44-220. Higher score indicates a higher level of mental pain. Change= (Day 15 score - baseline score).
Change from Day 15 in Orbach and Mikulincer Mental Pain scale (OMMPI) at Day 30. | Day 15 and Day 30.
  The experience of mental pain will be assessed using a self-report questionnaire (OMMPI; Orbach, Mikulincer, Sirota & Gilboa-Schechtman, 2003). The questionnaire contains 44 items. Each item is scored on a scale of 1-5, yielding a total score of between 44-220. Higher score indicates a higher level of mental pain. Change= (Day 30 score - Day 15 score).
Change from Baseline in Tolerance of Mental Pain Scale (TMPS) at Day 15. | Baseline and Day 15.
  The perceived ability of the individual to tolerate mental pain will be assessed using a self-report questionnaire (TMPS; Orbach, Gilboa-Schechtman, Johan, Mikulincer, 2004). The questionnaire contains 20 items. Each item is scored on a scale of 1-5, yielding a total score of between 20-100. Higher score indicates a greater perceived ability to tolerate mental pain. Change= (Day 15 score - baseline score).
Change from Day 15 in Tolerance of Mental Pain Scale (TMPS) at Day 30. | Day 15 and Day 30.
  The perceived ability of the individual to tolerate mental pain will be assessed using a self-report questionnaire (TMPS; Orbach, Gilboa-Schechtman, Johan, Mikulincer, 2004). The questionnaire contains 20 items. Each item is scored on a scale of 1-5, yielding a total score of between 20-100. Higher score indicates a greater perceived ability to tolerate mental pain. Change= (Day 30 score - Day 15 score).
Change from Baseline in Helplessness, Hopelessness, and Haplessness Scale (HHH) at Day 15. | Baseline and Day 15.
  Hopelessness and helplessness will be assessed by using a self-report questionnaire (Helplessness, Hopelessness, and Haplessness (HHH); Lester,2001). Originally the questionnaire contained three scales: hopelessness, helplessness, and haplessness. In the current study, only the hopelessness and helplessness scales will be used. Each scale contains 10 items, thus 20 items overall. Each item is scored between 1-6, yielding a total score of 20-120. Higher score indicates greater levels of hopelessness and helplessness. Change= (Day 15 score - baseline score).
Change from Day 15 in Helplessness, Hopelessness, and Haplessness Scale (HHH) at Day 30. | Day 15 and Day 30.
  Hopelessness and helplessness will be assessed by using a self-report questionnaire (Helplessness, Hopelessness, and Haplessness (HHH); Lester,2001). Originally the questionnaire contained three scales: hopelessness, helplessness, and haplessness. In the current study, only the hopelessness and helplessness scales will be used. Each scale contains 10 items, thus 20 items overall. Each item is scored between 1-6, yielding a total score of 20-120. Higher score indicates greater levels of hopelessness and helplessness. Change= (Day 30 score - Day 15 score).
Change from Baseline in Rosenberg Self-Esteem Scale (RSES) at Day 15. | Baseline and Day 15.
  Global self-esteem will be assessed using a self-report questionnaire (Rosenberg Self-Esteem Scale (RSES); Rosenberg, 1965). The questionnaire contains 10 items. Each item is scored on a scale of 1-4, yielding a total score of between 10-40. Higher score indicates higher levels of self-esteem. Change= (Day 15 score - baseline score).
Change from Day 15 in Rosenberg Self-Esteem Scale (RSES) at Day 30. | Day 15 and Day 30.
  Global self-esteem will be assessed using a self-report questionnaire (Rosenberg Self-Esteem Scale (RSES); Rosenberg, 1965). The questionnaire contains 10 items. Each item is scored on a scale of 1-4, yielding a total score of between 10-40. Higher score indicates higher levels of self-esteem. Change= (Day 30 score - Day 15 score).
Change from Baseline in Interpersonal Needs Questioner (INQ) at Day 15. | Baseline and Day 15.
  Interpersonal needs will be assessed using a self-report questionnaire (Interpersonal Needs Questioner (INQ); Van Orden, Cukrowicz, Witte, & Joiner, 2012). The questionnaire contains two scales: Perceived Burdensomeness (PB) and Thwarted Belongingness (TB). The scales contain 6 and 9 items, respectively. Each item is scored between 1-7, yielding a total score of 6-42 for PB, and 9-63 for TB. Higher scores indicate greater levels of perceived burdensomeness and thwarted belonging. Change= (Day 15 score - baseline score).
Change from Day 15 in Interpersonal Needs Questioner (INQ) at Day 30. | Day 15 and Day 30.
  Interpersonal needs will be assessed using a self-report questionnaire (Interpersonal Needs Questioner (INQ); Van Orden, Cukrowicz, Witte, & Joiner, 2012). The questionnaire contains two scales: Perceived Burdensomeness (PB) and Thwarted Belongingness (TB). The scales contain 6 and 9 items, respectively. Each item is scored between 1-7, yielding a total score of 6-42 for PB, and 9-63 for TB. Higher scores indicate greater levels of perceived burdensomeness and thwarted belonging. Change= (Day 30 score - Day 15 score).

SECONDARY OUTCOMES:
Change from Baseline in Cognitive Fusion Questionnaire (CFQ) at Day 15. | Baseline and Day 15.
  The extent to which a person is entangled in his thoughts and perceives them as unchangeable, will be assessed using a self-report questionnaire (Cognitive Fusion Questionnaire (CFQ); Gillanders et al., 2014). The questionnaire contains 7 items. Each item is scored on a scale of 1-7, yielding a total score of between 1-49. Higher score indicates greater levels of Cognitive fusion. Change= (Day 15 score - baseline score).
Change from Day 15 in Cognitive Fusion Questionnaire (CFQ) at Day 30. | Day 15 and Day 30.
  The extent to which a person is entangled in his thoughts and perceives them as unchangeable, will be assessed using a self-report questionnaire (Cognitive Fusion Questionnaire (CFQ); Gillanders et al., 2014). The questionnaire contains 7 items. Each item is scored on a scale of 1-7, yielding a total score of between 1-49. Higher score indicates greater levels of Cognitive fusion. Change= (Day 30 score - Day 15 score).

CONTACTS AND LOCATIONS:
Overall Officials: Sahak Yariv, Doctor, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreasson K, Krogh J, Bech P, Frandsen H, Buus N, Stanley B, Kerkhof A, Nordentoft M, Erlangsen A. MYPLAN -mobile phone application to manage crisis of persons at risk of suicide: study protocol for a randomized controlled trial. Trials. 2017 Apr 11;18(1):171. doi: 10.1186/s13063-017-1876-9. PMID 28399909
- [Background] Bhar S, Ghahramanlou-Holloway M, Brown G, Beck AT. Self-esteem and suicide ideation in psychiatric outpatients. Suicide Life Threat Behav. 2008 Oct;38(5):511-6. doi: 10.1521/suli.2008.38.5.511. PMID 19014303
- [Background] Allen NB. Cognitive therapy of depression. Aaron T Beck, A John Rush, Brian F Shaw, Gary Emery. New York: Guilford Press, 1979. Aust N Z J Psychiatry. 2002 Apr;36(2):275-8. doi: 10.1046/j.1440-1614.2002.t01-5-01015.x. No abstract available. PMID 11982561
- [Background] Beck AT, Brown G, Berchick RJ, Stewart BL, Steer RA. Relationship between hopelessness and ultimate suicide: a replication with psychiatric outpatients. Am J Psychiatry. 1990 Feb;147(2):190-5. doi: 10.1176/ajp.147.2.190. PMID 2278535
- [Background] Berk, M. S., Henriques, G. R., Warman, D. M., Brown, G. K., & Beck, A. T. (2004). A cognitive therapy intervention for suicide attempters: An overview of the treatment and case examples. Cognitive and Behavioral Practice, 11(3), 265-277.
- [Background] Brown GK, Beck AT, Steer RA, Grisham JR. Risk factors for suicide in psychiatric outpatients: a 20-year prospective study. J Consult Clin Psychol. 2000 Jun;68(3):371-7. PMID 10883553
- [Background] Brown GK, Ten Have T, Henriques GR, Xie SX, Hollander JE, Beck AT. Cognitive therapy for the prevention of suicide attempts: a randomized controlled trial. JAMA. 2005 Aug 3;294(5):563-70. doi: 10.1001/jama.294.5.563. PMID 16077050
- [Background] Chandrashekar P. Do mental health mobile apps work: evidence and recommendations for designing high-efficacy mental health mobile apps. Mhealth. 2018 Mar 23;4:6. doi: 10.21037/mhealth.2018.03.02. eCollection 2018. No abstract available. PMID 29682510
- [Background] Chu C, Buchman-Schmitt JM, Stanley IH, Hom MA, Tucker RP, Hagan CR, Rogers ML, Podlogar MC, Chiurliza B, Ringer FB, Michaels MS, Patros CHG, Joiner TE. The interpersonal theory of suicide: A systematic review and meta-analysis of a decade of cross-national research. Psychol Bull. 2017 Dec;143(12):1313-1345. doi: 10.1037/bul0000123. Epub 2017 Oct 26. PMID 29072480
- [Background] DeRubeis RJ, Hollon SD, Amsterdam JD, Shelton RC, Young PR, Salomon RM, O'Reardon JP, Lovett ML, Gladis MM, Brown LL, Gallop R. Cognitive therapy vs medications in the treatment of moderate to severe depression. Arch Gen Psychiatry. 2005 Apr;62(4):409-16. doi: 10.1001/archpsyc.62.4.409. PMID 15809408
- [Background] Ducasse D, Holden RR, Boyer L, Artero S, Calati R, Guillaume S, Courtet P, Olie E. Psychological Pain in Suicidality: A Meta-Analysis. J Clin Psychiatry. 2018 May/Jun;79(3):16r10732. doi: 10.4088/JCP.16r10732. PMID 28872267
- [Background] Ellis, T. E., & Rutherford, B. (2008). Cognition and Suicide: Two Decades of Progress. International Journal of Cognitive Therapy, 1(1), 47-68.
- [Background] Garlow SJ, Rosenberg J, Moore JD, Haas AP, Koestner B, Hendin H, Nemeroff CB. Depression, desperation, and suicidal ideation in college students: results from the American Foundation for Suicide Prevention College Screening Project at Emory University. Depress Anxiety. 2008;25(6):482-8. doi: 10.1002/da.20321. PMID 17559087
- [Background] Gillanders DT, Bolderston H, Bond FW, Dempster M, Flaxman PE, Campbell L, Kerr S, Tansey L, Noel P, Ferenbach C, Masley S, Roach L, Lloyd J, May L, Clarke S, Remington B. The development and initial validation of the cognitive fusion questionnaire. Behav Ther. 2014 Jan;45(1):83-101. doi: 10.1016/j.beth.2013.09.001. Epub 2013 Sep 18. PMID 24411117
- [Background] Jang JM, Park JI, Oh KY, Lee KH, Kim MS, Yoon MS, Ko SH, Cho HC, Chung YC. Predictors of suicidal ideation in a community sample: roles of anger, self-esteem, and depression. Psychiatry Res. 2014 Apr 30;216(1):74-81. doi: 10.1016/j.psychres.2013.12.054. Epub 2014 Jan 9. PMID 24507544
- [Background] Kohn R, Saxena S, Levav I, Saraceno B. The treatment gap in mental health care. Bull World Health Organ. 2004 Nov;82(11):858-66. Epub 2004 Dec 14. PMID 15640922
- [Background] Larsen ME, Nicholas J, Christensen H. A Systematic Assessment of Smartphone Tools for Suicide Prevention. PLoS One. 2016 Apr 13;11(4):e0152285. doi: 10.1371/journal.pone.0152285. eCollection 2016. PMID 27073900
- [Background] Lakey CE, Hirsch JK, Nelson LA, Nsamenang SA. Effects of contingent self-esteem on depressive symptoms and suicidal behavior. Death Stud. 2014 Jul-Dec;38(6-10):563-70. doi: 10.1080/07481187.2013.809035. Epub 2014 Feb 5. PMID 24499415
- [Background] Lester D. An inventory to measure helplessness, hopelessness, and haplessness. Psychol Rep. 2001 Dec;89(3):495-8. doi: 10.2466/pr0.2001.89.3.495. PMID 11824706
- [Background] Lester D. Defeat and entrapment as predictors of depression and suicidal ideation versus hopelessness and helplessness. Psychol Rep. 2012 Oct;111(2):498-501. doi: 10.2466/12.02.09.PR0.111.5.498-501. PMID 23234094
- [Background] Lester, D. (2012). The role of irrational thinking in suicidal behavior. Comprehensive Psychology, 1, 12-02.
- [Background] Orbach I, Mikulincer M, Sirota P, Gilboa-Schechtman E. Mental pain: a multidimensional operationalization and definition. Suicide Life Threat Behav. 2003 Fall;33(3):219-30. doi: 10.1521/suli.33.3.219.23219. PMID 14582833
- [Background] Orbach, I., Gilboa-Schechtman, E., Johan, M., Mikulincer, M., (2004). Tolerance for Mental Pain Scale. Bar-Ilan University, Ramat-Gan, Israel.
- [Background] Pauwels K, Aerts S, Muijzers E, De Jaegere E, van Heeringen K, Portzky G. BackUp: Development and evaluation of a smart-phone application for coping with suicidal crises. PLoS One. 2017 Jun 21;12(6):e0178144. doi: 10.1371/journal.pone.0178144. eCollection 2017. PMID 28636617
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Reynolds, W. (1991). ASIQ, adult suicidal ideation questionnaire: Professional manual. Psychological Assessment Resources, Incorporated.
- [Background] Roncero M, Belloch A, Doron G. Can Brief, Daily Training Using a Mobile App Help Change Maladaptive Beliefs? Crossover Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Feb 13;7(2):e11443. doi: 10.2196/11443. PMID 30758294
- [Background] Rosenberg, M. (1965). Rosenberg self-esteem scale (SES). Society and the adolescent self-image.
- [Background] Scott, A., & Guo, B. (2012). For which strategies of suicide prevention is there evidence of effectiveness. Denmark: World Health Organization.
- [Background] Shelef L, Fruchter E, Hassidim A, Zalsman G. Emotional regulation of mental pain as moderator of suicidal ideation in military settings. Eur Psychiatry. 2015 Sep;30(6):765-9. doi: 10.1016/j.eurpsy.2014.12.004. Epub 2015 Jun 29. PMID 26138045
- [Background] Stanley B, Brown G, Brent DA, Wells K, Poling K, Curry J, Kennard BD, Wagner A, Cwik MF, Klomek AB, Goldstein T, Vitiello B, Barnett S, Daniel S, Hughes J. Cognitive-behavioral therapy for suicide prevention (CBT-SP): treatment model, feasibility, and acceptability. J Am Acad Child Adolesc Psychiatry. 2009 Oct;48(10):1005-1013. doi: 10.1097/CHI.0b013e3181b5dbfe. PMID 19730273
- [Background] Tang TZ, DeRubeis RJ, Beberman R, Pham T. Cognitive changes, critical sessions, and sudden gains in cognitive-behavioral therapy for depression. J Consult Clin Psychol. 2005 Feb;73(1):168-72. doi: 10.1037/0022-006X.73.1.168. PMID 15709844
- [Background] Tighe J, Shand F, Ridani R, Mackinnon A, De La Mata N, Christensen H. Ibobbly mobile health intervention for suicide prevention in Australian Indigenous youth: a pilot randomised controlled trial. BMJ Open. 2017 Jan 27;7(1):e013518. doi: 10.1136/bmjopen-2016-013518. PMID 28132007
- [Background] Turecki G, Brent DA. Suicide and suicidal behaviour. Lancet. 2016 Mar 19;387(10024):1227-39. doi: 10.1016/S0140-6736(15)00234-2. Epub 2015 Sep 15. PMID 26385066
- [Background] Van Orden KA, Witte TK, Cukrowicz KC, Braithwaite SR, Selby EA, Joiner TE Jr. The interpersonal theory of suicide. Psychol Rev. 2010 Apr;117(2):575-600. doi: 10.1037/a0018697. PMID 20438238
- [Background] Van Orden KA, Cukrowicz KC, Witte TK, Joiner TE. Thwarted belongingness and perceived burdensomeness: construct validity and psychometric properties of the Interpersonal Needs Questionnaire. Psychol Assess. 2012 Mar;24(1):197-215. doi: 10.1037/a0025358. Epub 2011 Sep 19. PMID 21928908
- [Background] Verrocchio MC, Carrozzino D, Marchetti D, Andreasson K, Fulcheri M, Bech P. Mental Pain and Suicide: A Systematic Review of the Literature. Front Psychiatry. 2016 Jun 20;7:108. doi: 10.3389/fpsyt.2016.00108. eCollection 2016. PMID 27378956
- [Background] W.H.O. Preventing Suicide: A Global Imperative. Luxembourg: World Health Organization (2014).
- [Background] Witt K, Spittal MJ, Carter G, Pirkis J, Hetrick S, Currier D, Robinson J, Milner A. Effectiveness of online and mobile telephone applications ('apps') for the self-management of suicidal ideation and self-harm: a systematic review and meta-analysis. BMC Psychiatry. 2017 Aug 15;17(1):297. doi: 10.1186/s12888-017-1458-0. PMID 28810841
- [Background] Zalsman G, Hawton K, Wasserman D, van Heeringen K, Arensman E, Sarchiapone M, Carli V, Hoschl C, Barzilay R, Balazs J, Purebl G, Kahn JP, Saiz PA, Lipsicas CB, Bobes J, Cozman D, Hegerl U, Zohar J. Suicide prevention strategies revisited: 10-year systematic review. Lancet Psychiatry. 2016 Jul;3(7):646-59. doi: 10.1016/S2215-0366(16)30030-X. Epub 2016 Jun 8. PMID 27289303
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886